CLINICAL TRIAL: NCT04384666
Title: A Randomized, Open-Label, Crossover Study to Evaluate the Pharmacokinetic Profiles of Rotigotine After a Single Dose of LY03003 (28 mg) Versus After a Week of Daily NEUPRO® Transdermal Patch (4 mg Every 24 Hours) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LY03003/CT-USA-106
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Injections, Intramuscular; Injections; rotigotine

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, 2-sequence, 2-treatment cross-over study to evaluate the rotigotine PK profiles after a single dose of 28 mg LY03003 IM injection and 7 days of 4 mg NEUPRO® patch q24h in healthy subjects.
  Subjects will be screened according to the inclusion and exclusion criteria (Days -28 to -1) prior to randomization. Each subject will be randomized 1:1 to 1 of the 2 treatment sequences and will participate in 2 treatment periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY03003 (Experimental): LY03003 28 mg
  Interventions: Drug: LY03003 (rotigotine extended release microspheres for intramuscular [IM] injection)
- Neupro 4Mg/24Hr Transdermal Patch (Active Comparator): Neupro 4 mg / 24 Hr. Transdermal Patch
  Interventions: Other: Neupro 4 mg / 24 Hr. Transdermal Patch

INTERVENTIONS:
Drug: LY03003 (rotigotine extended release microspheres for intramuscular [IM] injection) — LY03003 (rotigotine extended release microspheres for intramuscular [IM] injection)
  Arms: LY03003
Other: Neupro 4 mg / 24 Hr. Transdermal Patch — Neupro 4 mg /24 Hr. Transdermal Patch
  Arms: Neupro 4Mg/24Hr Transdermal Patch

SUMMARY:
This is a randomized, open-label, 2-sequence, 2-treatment cross-over study in healthy adult subjects. Rotigotine PK profiles will be obtained from all subjects after both a single dose of 28 mg LY03003 and 1 week of 4 mg q24h NEUPRO® patch. Subjects will be randomized 1:1 to 1 of the 2 treatment sequences.

DETAILED DESCRIPTION:
Sequence 1

Period 1:

Subjects will check into the clinical research unit (CRU) on Day 0. On Day 1, subjects will receive the first 4 mg NEUPRO® patch in the morning. On Days 2 to 7, subjects will receive a 4- mg NEUPRO® patch every 24 hours (+/- 30 minutes) on one of the 7 designated patch application sites (see Section 12.2). On Day 1, serial PK samples will be collected within 30 minutes prior to patch application and 2, 4, 8, 12, 16, 20 hours post patch application. On Days 2, 3, 4, 5 and 6, one PK sample will be collected pre-patch (<30 minutes pre-patch) application only. On Day 7, the subjects will receive the NEUPRO® patch and serial PK samples will be collected pre-patch (<30 mins pre-patch) application and at 2, 4, 6, 8, 12, 16, 20, 24, 26, 28, 30, 33, 36, and 48 hours post-patch application Subject will stay at CRU till Day 14 to complete the End of Treatment ( EOT) procedures and prepare for the LY03003 treatment in Period 2 on the next day.

Period 2:

On Day 1 in the morning, subjects will receive a single-dose IM injection of 28 mg LY03003. Serial PK samples will be collected within 30 minutes pre-dosing and at 0.5, 1, 6, and 12 hours post dosing on Day 1. On Days 2 to Day 8, Day 10, Day 12, Day 15, Day 17, and Day 22, one single post-dose PK sample will be collected at the following corresponding hours: 24, 48, 72, 96, 120, 144, 168, 216, 264, 336, 384, and 504 hours post dosing. Subjects will stay at CRU till Day 22 to have PK collected and EOT activities completed. Subjects will be discharged on the same day. A 7-day safety follow-up period will be followed with a call on Day 29.

Sequence 2 Period 1 Subjects will check into the CRU on Day 0. In the morning of Day 1, subjects will receive a single-dose IM injection of 28 mg LY03003. Serial PK samples will be collected within 30 minutes pre-dosing and at 0.5, 1, 6 and 12 hours post dosing on Day 1. On Days 2 to Day 8, Day 10, Day 12, and Day 15, Day 17, and Day 22, one single postdose PK sample will be collected at the following corresponding hours: 24, 48, 72, 96, 120, 144, 168, 216, 264, 336, 384, and 504 hours post dosing. On Day 22, Subjects will have PK samples collected and EOT activities completed. Subjects will stay at the CRU until Day 29 and complete a 7-day washout period and to prepare for NEUPRO® patch treatment in Period 2 on the next day.

Period 2 On Day 1, subjects will receive the first 4 mg NEUPRO® patch in the morning. On Days 2 to 7, subjects will receive a 4- mg NEUPRO® patch every 24 hours (+/- 30 mins) on one of the 7 designated patch application sites (see Section 12.2). On Day 1, serial PK samples will be collected within 30 minutes prior to patch application and 2,4, 8, 12, 16 and 20 hours post patch application. On Days 2, 3, 4, 5 and 6, one PK sample will be collected pre-patch (<30 minutes pre-patch) application only. On Day 7, the subjects will receive the NEUPRO® patch and serial PK samples will be collected pre-patch (<30 minutes pre-patch) application and at 2, 4, 6, 8, 12, 16, 20, 24, 26, 28, 30, 33, 36, and 48 hours post-patch application. Subjects will stay at CRU and continue the safety follow-up period until Day14. On Day 14, subjects will complete EOT activities, followed by being discharged from the study on the same day.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of giving informed consent;
2. Between the ages of 18 and 45 years old, inclusive;
3. Healthy, per investigator's judgment, based on detailed medical history, clinical laboratory safety tests, vital signs, full physical examination, and ECG;
4. Nonsmoker defined as not having smoked or used any form of tobacco within 6 months before screening;
5. BMI between 18.5 and 30 kg/m2, inclusive, and body weight ≥50 kg at screening;
6. Willing and able to comply with study procedures, adhere to study restrictions, and stay at the CRU during in-subject stays required by the protocol;
7. All female subjects (childbearing potential and non-childbearing potential) must have a negative serum pregnancy test result at screening. In addition, female subjects must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion) based on subject report, or (iii) if of childbearing potential and heterosexually active, practicing or agree to practice a highly effective method of contraception. Highly effective methods of contraception include an intrauterine device (IUD), intrauterine hormone- releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable contraception method if the vasectomized partner is the sole sexual partner of the female subject and the vasectomized partner has received medical confirmation of surgical success. Highly effective methods of contraception must be used for at least 21 days prior to study drug dosing, throughout the study, and for another 90 days after the end of the study to minimize the risk of pregnancy.
8. All male subjects must be willing to use a condom in combination with another acceptable form of contraception (such as partner's use of a cap, diaphragm, sponge, spermicide, or hormonal contraception. Of note, male and female condom combination is NOT acceptable)during any sexual activity (e.g. vaginal, anal, oral) with women with childbearing potential (WOCBP) even if the subjects have undergone a successful vasectomy or if their partner is already pregnant or breastfeeding, from study drug dosing, throughout the study, and for another 90 days after the end of study.

Exclusion Criteria:

1. History of symptomatic orthostatic hypotension with a decrease of ≥20 mmHg in systolic blood pressure (SBP) or decrease of ≥10 mmHg in diastolic blood pressure (DBP) when changing from a supine to a standing position after having been in the supine position for at least 5 minutes or SBP less than 105 mmHg in a supine position at screening and Baseline;
2. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, and/or lipid metabolism disorders, and/or drug hypersensitivity;
3. History of epilepsy, seizures as an adult, lifetime history of stroke, or transient ischemic attack (TIA) within 1 year prior to screening and Baseline;
4. History of sleep attacks or narcolepsy;
5. Known or suspected malignancy within 5 years with the exception of treated and cured basal cell carcinoma (skin), squamous cell carcinoma (skin), or in-situ cervical carcinoma;
6. Positive blood screen for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
7. Positive pregnancy test result or plan to become pregnant if female;
8. Female who is pregnant or breastfeeding or of childbearing potential without adequate contraception (see Inclusion Criterion 7);
9. Hospital admission or major surgery within 30 days prior to screening and Baseline;
10. Receipt of another investigational product within one month or 5 half-lives of the other investigational product, whichever is longer, before study drug administration in this study.
11. Presence of ink tattoos of any kind in any of the designated patch application sites.
12. History of prescription drug abuse or any illicit drug use within 6 months prior to screening and Baseline;
13. History of alcohol abuse according to medical history within 6 months prior to screening and Baseline;
14. Positive screen for alcohol, drugs of abuse and cotinine;
15. Unwillingness or inability to comply with food and beverage restrictions during study participation;
16. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening and Baseline;
17. Use of prescription or over-the-counter (OTC) medications and/or herbal supplements (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3 g/day is permitted until 24 hours prior to dosing);
18. Inability to tolerate study drug in any prior rotigotine or LY03003 trial or intolerance or hypersensitivity to rotigotine or any excipients or diluents (Poly (lactide-co-glycolide) [PLGA], carboxymethylcellulose sodium [SCMC], stearic acid, or mannitol);
19. History of known intolerance/hypersensitivity to antiemetics such as ondansetron, tropisetron, and glycopyrrolate;
20. History of suicide attempt in the past 6 months and/or seen by the investigator as having a significant history of risk of suicide or homicide;
21. Unwillingness of male participants to use appropriate contraceptive measures (see Inclusion Criteria 8) if engaging in sexual intercourse with a female partner of childbearing potential throughout the study and for at least 1 month after the end of the study, plus an additional 60 days.
22. Unwillingness to refrain from sexual intercourse with pregnant or lactating women throughout the study and for at least 1 month after the end of the study;
23. Any other clinically relevant hepatic, renal, hematologic, and/or cardiac dysfunction, or other medical condition, or clinically significant laboratory abnormality that would interfere with the subject's safety or study outcome in the judgment of the investigator.
24. A lifetime history of bipolar I disorder, bipolar II disorder, cyclothymia or other specified bipolar and related disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 34 days

SECONDARY OUTCOMES:
Adverse Events | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Sabet, MD, Principal Investigator — Pharmaceutical Research Associates
Locations (1):
- Pharmaceutical Research Associates, Inc., Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No